CLINICAL TRIAL: NCT04869462
Title: Prospective, Monocentric, Single Arm, Observational PMCF - Study on the Performance and Safety of Double-Shank Titanium Ligation Clip in Urology (Prostatectomy and Nephrectomy)
Brief Title: DS Titanium Ligation Clip in Urology (Prostatectomy and Nephrectomy)
Acronym: DOSTILCU
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2041
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer; Kidney Cancer; Congenital Abnormality of Kidney; Nephrolithiasis; Kidney Tuberculosis; Nephritis; Kidney Injury; Hydronephrosis
Keywords: Ligature of vessels and hollow organs; Marking of anatomic structures for radiological detection; Ligation; Prostatectomy; Nephrectomy; Minimally Invasive Surgical Procedures; Laparoscopy
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Nephrolithiasis; Tuberculosis, Renal; Nephritis; Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, monocentric, single arm, observational PMCF - Study on the Performance and Safety of Double-Shank Titanium Ligation Clip in Urology (Prostatectomy and Nephrectomy)

DETAILED DESCRIPTION:
The objective of this observational study is to collect systematically and proactively data regarding the Aesculap® DS Titanium Ligation Clip under daily clinical practice when used in urology in different indications.

The hypothesis of this study is that this event, slippage / movement of the clip, is extremely rare through the design if used in accordance with the Instructions for Use (IfU). The observed rate through the total number of clips might be a valuable parameter and could influence future research.

Furthermore, this study is one of the PMCF measures which enable the manufacturer to monitor the safety and performance of the Aesculap® DS Titanium Ligation Clips. The products bear the CE-marking and are routinely used within this institution for the above-mentioned procedures.

ELIGIBILITY:
Inclusion: Inclusion Criteria:

* Planned Da Vinci radical prostatectomy using DS Titanium Ligation Clips (according to the IfU) - OR
* Planned laparoscopic nephrectomy using Titanium Ligation Clip (according to the IfU) - OR
* Planned Da Vinci partial nephrectomy using Titanium Ligation Clip (according to the IfU)
* Patient's written informed consent
* Age ≥ 18 years
* Intraoperative Usage of DS Titanium Ligation Clips (according to the IfU)

Exclusion: Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data is collected preoperatively, intraoperatively and until discharge of all consecutive patients fulfilling the inclusion and exclusion criteria in a single site.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Rate of slippage / movement of the clip in relationship to the total number of used clips. | Intraoperatively
  Slippage / movement of the Aesculap® DS Titanium Ligation Clip is an observable slippage, movement, or rotation after the clip was successfully applied and the application forceps was removed. The number of observed slippage / movement of the clip will be documented on the CRF, the clip size, step of the procedure and further measures were necessary, i.e. removal of the clip or application of another clip, will be documented.
  In the end the rate will be brought in relationship to the overall number of applied clips. Thus, the number of applied clips is documented, for each clip size.

SECONDARY OUTCOMES:
Rate of Adverse events (intra- and postoperative) | up to discharge from hospital (approximately 10 days post surgery)
  * Postoperative bleedings
  * Infections
  * Urine extravasation in partial nephrectomy
  * Prolonged urinary catheter drainage in radical prostatectomies
  * Ileus
  * Venous thrombo-embolic events
  * Sepsis
  * Other

OTHER OUTCOMES:
intraoperative blood loss | intraoperatively
  Estimated intraoperative blood loss
Total operative time | intraoperatively
  Estimated operative time from first cut to last stitch
Length of hospital stay | up to discharge from hospital (approximately 10 days post surgery)
  Length of patient's stay in hospital after surgery
Handling parameters | intraoperatively
  The handling performance of the clip is assessed on a five point likert scale (very good, good, acceptable, poor) in four different handling aspects

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Simon, PD Dr. med., Principal Investigator — Ortenau KlinikumKlinik für Urologie und Kinderurologie ChefarztEbertplatz 1277654 Offenburg
Locations (1):
- Ortenau Klinikum Klinik für Urologie und Kinderurologie, Offenburg, Germany